CLINICAL TRIAL: NCT05140252
Title: Avoiding Low-value Treatments in Older Women With Early-stage Breast Cancer: Piloting a Patient Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2021.087; HUM00195321 (Other: University of Michigan)
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: de-implementation strategies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer decision aid (Experimental): Participants receive a breast cancer decision aid.
  Interventions: Behavioral: Breast cancer decision aid

INTERVENTIONS:
Behavioral: Breast cancer decision aid — The decision aid is tailored from a previously published aid, specific to women ≥70 with early-stage breast cancer. The aid will be delivered via mail or electronically per patient preference before the patient's initial appointment with a surgeon.

SUMMARY:
The aim of this study is to learn whether participants find a patient guide to breast cancer treatment decisions acceptable and appropriate for use.

DETAILED DESCRIPTION:
This study seeks to adapt and pilot test de-implementation strategies targeting low-value breast cancer treatments which have persisted despite national recommendations. Breast cancer is an ideal setting in which to study de-implementation given it is common, well-studied, typically presents at an early-stage, and care is provided primarily in a community setting.

ELIGIBILITY:
Inclusion Criteria

* Early stage breast cancer that is hormone receptor positive (HR+) and human epidermal growth factor negative (HER2-)
* Meet criteria for omission of sentinel lymph node biopsy (SLNB)
* Receiving care at Michigan Medicine

Exclusion Criteria

* Non-English speaking
* Male patients (current data does not support omission of SLNB in men)

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention (AIM) Survey | 1 week after receiving decision aid
  AIM is a validated, 4-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.
Intervention Appropriateness Measure (IAM) | 1 week after receiving decision aid
  IAM is a validated, 4-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.
Engagement with the patient decision aid | 1 week after receiving decision aid
  To determine feasibility, participants will be asked whether they engaged with the patient decision aid (1=thoroughly, 2=somewhat or 3=not at all), scored as a mean. The median score across all participants will be reported.

SECONDARY OUTCOMES:
Satisfaction with decision (SWD) | up to 120-days following surgery
  The SWD survey will be administered by telephone between 60- and 120-days following surgery. SWD is a validated, 6-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.
Treatment choice | 90 days after surgery
  The research team will access participants electronic medical records to determine the number of participants who underwent SLNB, radiation treatment, both or neither after surgery. This will be reported in 4 categories: Only SLNB, Only Radiation, Both or Neither.

CONTACTS AND LOCATIONS:
Overall Officials: Lesly A Dossett, MD, MPH, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schonberg MA, Freedman RA, Recht AR, Jacobson AR, Aliberti GM, Karamourtopoulos M, Nakhlis F, McCarthy EP, Pories SE, Sharma R, Dominici LS. Developing a patient decision aid for women aged 70 and older with early stage, estrogen receptor positive, HER2 negative, breast cancer. J Geriatr Oncol. 2019 Nov;10(6):980-986. doi: 10.1016/j.jgo.2019.05.004. Epub 2019 May 24. PMID 31130442